CLINICAL TRIAL: NCT01400763
Title: Bioavailability of Lutein From a Lutein-enriched Egg-yolk-beverage and Its Dried Re-suspended Versions.
Brief Title: Lutein Bioavailability From Fresh and Dried Beverages
Acronym: METC-11/07
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Meike Bunger, Wageningen University and Research Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EYEPOWDER
Record Dates: First submitted 2011-07-20; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Macular Pigment
Keywords: focus of study

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Fresh lutein-enriched egg-yolk beverage — Fresh lutein-enriched egg-yolk beverage
  Other Names: NWT-02
Dietary Supplement: Dried-1 lutein-enriched egg-yolk beverage — Dried-1 lutein-enriched egg-yolk beverage
Dietary Supplement: Dried-2 lutein-enriched egg-yolk beverage — Dried-2 lutein-enriched egg-yolk beverage
Dietary Supplement: Placebo beverage — Placebo beverage

SUMMARY:
Macular pigment is composed primarily of the xanthophylls lutein and zeaxanthin, which are members of the carotenoid family. Epidemiological evidence indicates that a higher intake of lutein and zeaxanthin is associated with a lower risk to develop age-related macular degeneration (AMD). The lipid matrix of an egg yolk is an excellent vehicle for the efficient absorption of dietary lutein and it is possible to increase the natural lutein concentration in an egg yolk. A fresh lutein-enriched egg yolk beverage has been produced using these lutein-enriched egg-yolks. However, this beverage has a limited shelf life of maximum three weeks. Drying this fresh beverage extents the shelf live, however, this should be without loosing its functional properties concerning lutein bioavailability. At WUR-FBR two types of drying procedures have been evaluated resulting in two different dried product formulations, which need to be tested. The question is, whether the lutein bioavailability is not affected by different drying procedures.

ELIGIBILITY:
Inclusion Criteria:

* age 18-35 years
* BMI 18-25 kg/m2
* body weight should be stable for ≥6 months (with no weight gain/loss > 3 kg)

Exclusion Criteria:

* use of medication except incidental use of pain killers
* pulmonary inhalation medication and except usage of the contraceptive pill
* chronic diseases such as IBD or other stomach or bowel diseases
* not willing to discontinue consumption of vitamin supplements
* allergic to cow milk / dairy products/ eggs/ egg-rich products
* vegetarians
* smoking
* pregnant or breastfeeding women
* having donated blood (as blood donor) within 1 month prior to the screening
* visit or planning to do so during the study
* impossible or difficult venapuncture

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Serum lutein concentration | six weeks after intervention

SECONDARY OUTCOMES:
Serum lipid concentrations | six weeks after intervention